CLINICAL TRIAL: NCT04770038
Title: Social Integration During Psychiatric Inpatient Therapy as Predictor of Treatment Response
Acronym: SANITY
Status: Completed | Type: Observational
Sponsor: University of Oldenburg (Other)
Collaborators: Prof. René Hurlemann (Unknown); Jella Voelter, M.Sc. (Unknown)
Responsible Party: Principal Investigator, Dirk Scheele, Prof., Ruhr University of Bochum
Other Study IDs: SANITY
Record Dates: First submitted 2021-02-04; First posted 2021-02-25 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: social integration; Borderline Personality Disorder; treatment response; psychiatric inpatient treatment; fMRI; negative social bias; social touch; interoception; trust; Dialectical Behavior Therapy
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples to measure cortisol, oxytocin and alpha-amylase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: 56 BPD patients
  Interventions: Behavioral: Dialectical Behavior Therapy (DBT)
- Control Group: 31 Healthy participants

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy (DBT) — Evidence-based psychotherapy for the treatment of Borderline Personality Disorder
  Groups: Patient Group

SUMMARY:
The present longitudinal study aims at (i) identifying neurobiological mechanisms associated with successful social integration during the treatment of inpatients with Borderline Personality Disorder (BPD) and (ii) improving biomarker-based predictions of treatment response by incorporating core metrics of social integration.

DETAILED DESCRIPTION:
Social connections have a strong impact on mental and physical health. Surprisingly, however, there is a paucity of studies probing the predictive validity of perceived social connections such as subjective social support and loneliness for the outcomes of inpatient treatment of BPD. Although social impairments are key features of BPD psychopathology, social integration has been largely neglected, which may therefore explain the minimal translation of predictive molecular or imaging-based biomarkers into the clinic. The investigators hypothesize that the assessment of negative cognitive biases at baseline will help to identify BPD patients who will experience less social support and more loneliness during inpatient treatment. Furthermore, an inclusion of social integration indices may increase the incremental validity for the biomarker-based prediction of treatment response.

In this longitudinal, observational study, data from 56 BPD patients will be analyzed to assess negative cognitive biases and the underlying neurobiological mechanisms with behavioral, neuroendocrine, psychophysiological, and neural readouts before and after one month of inpatient Dialectical Behavior Therapy (DBT). To evaluate pathological biases, the patients' data will be compared with a control group of 31 healthy participants who will also be tested twice. Neural readouts include structural and functional magnetic resonance imaging (fMRI) measurements. The fMRI tasks will probe the processing of social touch, interpersonal trust, and interoception. To further investigate pathological distortions of social touch and interoception, interoceptive accuracy and comfort zones of social touch will be assessed. Further, patients and healthy participants will perform a positive social interaction task, accompanied by psychophysiological and neuroendocrinological measures. Psychometric questionnaires and semi-structured interviews will be used to monitor symptom load and social indices before, during, and after the inpatient treatment. Long-term effects will be assessed by questionnaires and interviews 8 and 20 weeks after inpatient treatment/waiting time, as well as after each DBT module (follow-ups). The investigators plan to conduct uni- and multivariate analyses of the baseline measurements to predict patients' social integration and treatment response during the inpatient therapy and examine treatment-related changes. The findings of this project may help identify vulnerable patients that benefit from adjunct therapies targeting negative social biases and improve biomarker-based models of treatment prediction.

ELIGIBILITY:
Inclusion Criteria:

* Willingness / ability to give written informed consent to participate in the study
* BPD patients: on a waiting list for DBT, BPD as primary diagnosis
* Healthy participants: free of current physical or psychiatric illness
* Fluent in German

Exclusion Criteria:

* Contraindication for MRI investigation (e.g. agoraphobia, pacemaker, pregnancy)
* Acute suicidality, current substance dependence or primary psychotic disorder
* A history of head trauma or neurological illness
* Scars on a predefined skin area (approx. 20 cm) of the shins
* Healthy participants: current or past psychiatric inpatient treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: BPD patients are recruited from a waiting list for DBT inpatient treatment and directly during inpatient treatment at the University Clinic for Psychiatry and Psychotherapy, Karl-Jaspers-Klinik, Bad Zwischenahn, Germany.
  Group 2: Healthy participants are recruited via the notice board of the University of Oldenburg, and, in order to achieve a more heterogenous sample, via online advertisments
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Social integration during inpatient treatment as measured by questionnaires and interviews | Social integration (duration approx. 30-45 minutes) will be measured continuously during inpatient treatment (twice a week for four weeks).
  Social integration will be assessed with questionnaires and interviews (e.g. the perceived social support questionnaire).
Changes in neural responses to interpersonal touch | The fMRI task (duration approx. 15 minutes) will be performed before and after one month of inpatient DBT/waiting time.
  Blood-oxygen-level-dependent (BOLD) signal will be assessed while participants undergo a social touch task. Conditions consist of four types of touch trials with combinations of slow (~ 5 cm/s) and fast touch (~ 20 cm/s), as well as social (administered by hand) and non-social (administered with a brush) touch and a control (no touch) condition. An experimenter, who cannot be seen by the participant, will administer the touch across 20 cm of the shins. After each trial, participants will be asked to rate how comforting the touch was perceived. The neural responses to interpersonal touch will be compared before and after DBT-treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in comfort ratings of interpersonal touch in the fMRI task | The fMRI task (duration approx. 15 minutes) will be performed before and after one month of inpatient DBT/waiting time.
  During the social touch fMRI task, participants rate the comfort of the trial on a Visual Analogue Scale (VAS). The behavioral data will be analyzed and linked to the BOLD signal. Comfort ratings will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in neural responses in the Trust Game | The fMRI task (duration approx. 6 minutes) will be performed before and after one month of inpatient DBT/waiting time.
  BOLD signal will be measured while participants play a single-round trust game in the role of an investor. Participants will have to decide how much money they want to invest in an unknown trustee without receiving feedback about the decisions of the trustees. In a control condition, participants will play a risk game and invest money in a computer, which will randomly decide whether the money will be shared. The neural correlates will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in interpersonal trust | The fMRI task (duration approx. 6 minutes) will be performed before and after one month of inpatient DBT /waiting time.
  During the fMRI Trust Game, participants will decide how much (from 1 Euro to 10 Euro) they want to invest in the unknown trustees on a VAS. Furthermore, participants will rate the facial trustworthiness of the face stimuli used in the fMRI Trust Game. These behavioral data will be analyzed and linked to the BOLD signal. The behavioral data will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in neural responses during an interoception task | The fMRI task (duration approx. 13 minutes) will be performed before and after one month of inpatient DBT/waiting time.
  During the interoception fMRI task, participants are instructed to focus on their heart, their stomach, or color changes of the word "target" (as control). After every second trial, participants rate how intensely they perceived their heart or their stomach. During the control condition, participants indicate how intensely they perceived the color change. The neural correlates will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in intensity ratings of bodily awareness in the fMRI task | The fMRI task (duration approx. 13 minutes) will be performed before and after one month of inpatient DBT/waiting time.
  During the interoception fMRI task, participants rate how intensely they perceived their heart or their stomach on VAS. The behavioral data will be analyzed and linked to the BOLD signal. Intensity ratings will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in interoceptive accuracy as measured by a heartbeat discrimination task | Interoceptive accuracy (duration approx. 20 minutes) will be assessed before and after one month of inpatient DBT/waiting time.
  During the heartbeat discrimination task, participants have to indicate, whether a series of tones is presented synchronously or asynchronously to their own heartbeat. In addition, they rate their confidence on their own assessment on a VAS. Interoceptive accuracy will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in interoceptive sensibility as measured with a questionnaire | Interoceptive sensibility (duration approx. 5 minutes) will be measured before and after one month of inpatient DBT/waiting time.
  The Multidimensional Assessment of Interoceptive Awareness (MAIA-2) will be used to measure self-reported interoceptive sensibility. Questionnaire scores will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in psychophysiological measures during a positive social interaction | The positive social interaction (duration approx. 15 minutes) will be conducted before one month of inpatient DBT/waiting time
  The positive social interaction will consist of a semi-structured ten-minute conversation between the participant and a same-sex unfamiliar experimenter. After a baseline measurement of five minutes, participants will talk about plans for a fictive lottery win and hobbies and interests. During the baseline, as well as during the conversation, psychophysiological parameters of both, the participant and the experimenter, will be measured simultaneously.
Changes in hormone and enzyme salivary concentrations in response to a positive social interaction | The positive social interaction (duration approx. 15 minutes) will be conducted before one month of inpatient DBT/waiting time
  Saliva samples will be collected before, immediately after, and 15 minutes after the social interaction task.
Changes in mood in response to a social interaction | The positive social interaction (duration approx. 15 minutes) will be conducted before one month of inpatient DBT/waiting time
  Mood state will be assessed with questionnaires (e.g. the Profile of Mood States (POMS)).
Changes in bodily maps of social touch | The bodily maps (duration approx. 10-15 minutes) will be assessed before and after 4-weeks DBT treatment/waiting time.
  In a computerized task, participants will indicate on a human silhouette, where a specific person (e.g. their mother) would be allowed to touch them in everyday situations. Comfort zones of social touch for different members of their social network (e.g. brother, female stranger etc.) will be analyzed. Bodily maps will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in attitude towards social touch | Self-reported touch preferences (duration approx. 5 minutes) will be assessed before and after one month of inpatient DBT/waiting time as well as during follow-up measurements.
  The attitude towards social touch will be measured by the Social Touch Questionnaire (STQ). Self-reported touch preferences will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in negative social biases | Questionnaires (duration approx. 15-20 minutes) will be measured before and after one month of inpatient DBT/waiting time as well as during follow-up measurements.
  Negative social biases will be assessed with questionnaires (e.g. the University of California Los Angeles (UCLA) Loneliness Scale). Questionnaire scores will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in symptom load | Symptom load (duration approx. 30-45 minutes) will be measured before and after one month of inpatient DBT, continuously during therapy (twice a week for four weeks) as well as during follow-up measurements.
  Symptom load will be assessed with questionnaires and interviews (e.g. the Borderline-Symptom-List-23 (BSL-23)). Symptom load will be compared before and after the DBT treatment and will be measured continuously during DBT treatment.

SECONDARY OUTCOMES:
Changes in neural activity at resting state | Resting State (duration approx. 10 minutes) will be performed before and after one month of inpatient DBT/waiting time.
  fMRI will be performed to measure BOLD-signal while participants lay in the MRI-scanner with eyes open. Participants will be instructed to look at a fixation cross for ~ 10 minutes. The neural correlates will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in vigilance | Vigilance (duration approx. 5 minutes) will be measured one week before and after one month of inptatient DBT/waiting time.
  Vigilance will measured with the Psychomotor Vigilance Task (PVT). The PVT is a reaction time task in which participants respond to visual stimuli via button presses. Participants fixate a black screen and press a button as soon as a digital clock with a running time-measurement appears on screen. Vigilance will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Childhood maltreatment | The CTQ (duration approx. 5 minutes) will be performed before one month of inpatient DBT/waiting time.
  The Childhood Trauma Questionnaire (CTQ) will be used to measure childhood maltreatment. The scale ranges between 5 and 100 points and higher scores indicate higher childhood maltreatment.
Changes in symptom load of possible comorbidities | Symptom load (duration approx. 10 minutes) will be measured before and after one month of inpatient DBT treatment/waiting time as well as during follow-up measurements.
  Symptom load will be assessed with questionnaires (e.g. the Becks-Depression-Inventory-II (BDI-II)). Questionnaire scores will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Changes in personality traits | Personality traits (duration approx. 10 minutes) will be measured before and after one month of inpatient DBT/waiting time.
  The big five personality traits will be measured with the NEO-Five-Factor-Inventory (NEO-FFI). Personality traits will be compared before and after the DBT treatment and the treatment-induced changes will be compared with changes in the healthy control group.
Psychotherapy outcome as measured with a questionnaire | Psychotherapy outcome (duration approx. 5 minutes) will be measured after one month of inpatient DBT.
  Psychotherapy outcome will be assessed with the Bochum Change Questionnaire 2000 (BCQ-2000).
Verbal intelligence | Verbal intelligence (duration approx. 5 minutes) will be measured before one month of inpatient DBT/waiting time.
  Verbal intelligence will be measured with the Multiple Choice Vocabulary Test (MWT-B).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Scheele, Prof., Principal Investigator — Ruhr University of Bochum, Germany
Locations (1):
- Department of Psychiatry, University of Oldenburg, Karl-Jaspers-Klinik, Bad Zwischenahn, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Research group website — http://www.dirk-scheele.org
- See also: Research group website — http://www.hurlemannlab.com/